CLINICAL TRIAL: NCT04940845
Title: A Randomized, Single-blinded and Parallel Study to Assess the Pharmacokinetic, Safety and Immunogenicity of HS-20090-2 Injection and Prolia® in Healthy Adults
Brief Title: Comparing of the Pharmacokinetic, Safety and Immunogenicity of HS-20090-2 Injection and Prolia® in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Hansoh Biomedical Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Hansoh BioMedical R&D Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HS-20090-2-101
Record Dates: First submitted 2021-06-24; First posted 2021-06-28 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Postmenopausal Osteoporosis
Keywords: osteoporosis，postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-20090-2 (Experimental)
  Interventions: Drug: HS-20090-2
- Prolia® (Active Comparator)
  Interventions: Drug: Prolia

INTERVENTIONS:
Drug: HS-20090-2 — Subcutaneously injection of HS-20090-2 (60mg/1mL) once on the first day
  Arms: HS-20090-2
Drug: Prolia — Subcutaneously injection of Prolia® (60mg/1mL) once on the first day
  Arms: Prolia®

SUMMARY:
A randomized, single-blind and parallel group study to compare the pharmacokinetic, safety and immunogenicity of HS-20090-2 60mg#1ml#and Prolia® in healthy adults.

DETAILED DESCRIPTION:
This is a phase I, single center, randomized, single-blind and parallel group clinical trial .The primary objective is to assess the pharmacokinetic similarity of single subcutaneously injection of HS-20090-2 or Prolia® in healthy volunteers.The secondary objectives are to assess the Clinical safety and immunogenicity similarity of single subcutaneously injection of HS-20090-2 or Prolia® in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form and fully understand the test content, process and possible adverse reactions, and be able to complete the study according to the test plan requirements;
2. Healthy males, Aged ≥18 years or ≤50 years old(including the boundary value);
3. Agree to take effective contraceptive measures throughout the study period until at least 6 months after the last drug is administered;
4. Clinical laboratory examination, chest X-ray, abdominal B-ultrasound, electrocardiogram, physical examination, vital signs and various examinations are normal or abnormal without clinical significance.

Exclusion Criteria:

1. Occurred or suffering from osteomyelitis or ONJ (mandibular necrosis) previously; The dental or jaw disease that is active, requiring oral surgery; or planned for invasive dental surgery during the study; or dental or oral surgery wounds have not healed;
2. Serum calcium levels are outside the normal range of the laboratory.
3. Subject has positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result viral hepatitis (including hepatitis B and hepatitis C), or positive HIV antibodies, or positive test for syphilis.
4. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 3 months or 5 half-lives (whichever is longer).
5. Prior use of medications within 12 months before and during the study. This includes medications such as, but not limited to: Bisphosphonates Fluoride Calcitonin Strontium Parathyroid hormone or derivatives Supplemental vitamin D (>1000 IU/day) Glucocorticosteroids (topical corticosteroids administered more than 2 weeks prior to enrolment are allowed) Anabolic steroids Calcitriol Diuretics

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-infinity curve (AUC0-∞ ) | 155days
  Area under the plasma concentration-time curve (AUC0-t ) from 0 o'clock to infinite time.
Cmax | 155days
  maximum concentration

SECONDARY OUTCOMES:
Adverse events(AE) | 155days
  The adverse medical events that occur after the clinical trial subjects receive the test drug do not necessarily have a causal relationship with the treatment.
ADA | 155days
  percentage of subjects positive for antidrug antibody
Nab | 155days
  percentage of subjects positive for Nab

CONTACTS AND LOCATIONS:
Overall Officials: Dong Liu, PhD, Principal Investigator — Huazhong University of Science and Technoogy; Xiuhua Ren, Master, Principal Investigator — Huazhong University of Science and Technoogy
Locations (1):
- Huazhong University of Science and Technoogy, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No